CLINICAL TRIAL: NCT06123780
Title: Pattern of Micro-bacterial Infection and Its Sensitivity to Antibiotics in COPD Patients With Acute Exacerbation.
Brief Title: Pattern of Microbial Infection in AECOPD Patients and Its Sensitivity to Antibiotics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Nazif Abdel-Tawab Mousa, Assistant lecturer, Assiut University
Other Study IDs: Bacteriology in AECOPD
Record Dates: First submitted 2023-10-11; First posted 2023-11-09 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Acute Exacerbation COPD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Measurement of bacterial species causing AECOPD and their Sensitivity pattern to antibiotics.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a major cause of chronic morbidity and mortality worldwide.

Acute exacerbation is a common problem during the natural course of COPD, which is characterized by an increase in the patient's daily symptoms of dyspnea, cough, and/or sputum beyond normal day-to-day variability and severe enough to require an additional therapy.

The most common cause of acute exacerbations of COPD (AECOPD) is an infection of the tracheobronchial tree and air pollution. As many as one-third of AECOPD causes are never identified. The microbial aetiology of AECOPD includes bacteria and viruses with more than 50% of cases being caused by bacterial infection.

The bacterial etiologies of AECOPD keep changing from time to time and the choice of antimicrobial depends upon on local prevalence of bacterial etiologies and their resistance pattern.

Antibiotics are the main form of treatment for AECOPD which are often initiated empirically based on healthcare provider's previous experiences , which often lead to the inappropriate use of antibiotics , thereby contributing to Antimicrobial Resistance.

Early diagnosis and knowledge of the predominant bacterial etiologies and antimicrobial resistance patterns will also help to correct treatment protocol for the management of AECOPD.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age and less than 80 years of age for both genders
* Confirmed diagnosis of COPD by spirometry
* Must be an AECOPD patient (with increased grade of dyspnea, increased purulence and amount of sputum) and admitted to the chest department or ICU
* Positive sputum culture

Exclusion Criteria:

* Age less than 18 years old
* Any associated pulmonary co-morbidity

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Demographic characteristics of these patients will be recorded, including sex, age, smoking status, underlying comorbidities, occupation and number of exacerbations.
  Clinical features will be recorded including increase grade of dyspnea , purulence and amount of sputum , history of previous NIV or MV.
  Spirometry as a confirmation tool of COPD. Arterial blood gases on admission. Complete blood count ( CBC ) and ESR Radiological profile of COPD patients. Sputum sample ; Spontaneous sputum sample by asking the patient to cough up sputum into sterile container.
  NIV patients : by spontaneous sputum sample. MV patients : by sputum suction through the endotracheal tube .
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Pattern of Microbial infection based on sputum culture results. | Baseline
  Identification of causative Microbial organisms of AECOPD based on results of sputum culture.
Pattern of antimicrobial sensitivities based on sputum culture results. | Baseline
  Identification of antimicrobial sensitivities and resistance patterns in this population based on results of sputum culture.

SECONDARY OUTCOMES:
Hospital length of stay | Baseline
  Exploring the relationship between the different causative organisms of AECOPD and the hospital length of stay.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled H. Ahmed, Professor, Study Director — Assuit U; Samiaa H Sadek, Professor, Study Director — Assuit U

REFERENCES:
- [Background] Venkatesan P. GOLD report: 2022 update. Lancet Respir Med. 2022 Feb;10(2):e20. doi: 10.1016/S2213-2600(21)00561-0. Epub 2021 Dec 20. No abstract available. PMID 34942084
- [Background] Rodriguez-Roisin R. Toward a consensus definition for COPD exacerbations. Chest. 2000 May;117(5 Suppl 2):398S-401S. doi: 10.1378/chest.117.5_suppl_2.398s. PMID 10843984
- [Background] Sethi S, Murphy TF. Infection in the pathogenesis and course of chronic obstructive pulmonary disease. N Engl J Med. 2008 Nov 27;359(22):2355-65. doi: 10.1056/NEJMra0800353. No abstract available. PMID 19038881
- [Background] Momanyi L, Opanga S, Nyamu D, Oluka M, Kurdi A, Godman B. Antibiotic Prescribing Patterns at a Leading Referral Hospital in Kenya: A Point Prevalence Survey. J Res Pharm Pract. 2019 Oct 16;8(3):149-154. doi: 10.4103/jrpp.JRPP_18_68. eCollection 2019 Jul-Sep. PMID 31728346
- [Background] Slone DE, Ganjam VK, Purohit RC, Ravis WR. Cortisol (hydrocortisone) disappearance rate and pathophysiologic changes after bilateral adrenalectomy in equids. Am J Vet Res. 1983 Feb;44(2):276-9. PMID 6830017